CLINICAL TRIAL: NCT04698850
Title: Brolucizumab vs. Aflibercept for Retinal Angiomatous Proliferation - Prospective Randomised Study
Brief Title: Brolucizumab vs. Aflibercept for Retinal Angiomatous Proliferation
Acronym: BEY-RAP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding issues
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Martin Pencak, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEY-RAP V1.0
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Wet Macular Degeneration
Keywords: wet age-related macular degeneration; retinal angiomatous proliferation; aflibercept; brolucizumab
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aflibercept (Active Comparator): Patients with RAP who will be receiving aflibercept.
  Interventions: Drug: Aflibercept 40 MG/ML [Eylea]; Drug: Ranibizumab 6 MG/ML [Lucentis]
- brolucizumab (Experimental): Patients with RAP who will be receiving brolucizumab.
  Interventions: Drug: Brolucizumab-Dbll 120 MG/ML [Beovu]; Drug: Ranibizumab 6 MG/ML [Lucentis]

INTERVENTIONS:
Drug: Aflibercept 40 MG/ML [Eylea] — Patients will be receiving intravitreal aflibercept starting with 3 monthly doses and continuing with treat-and-extend regimen with minimal interval of 8 week and maximum interval of 16 week. Interval can be prolonged or shortened by 2 or 4 weeks based on the disease activity and BCVA..
  Other Names: Eylea
  Arms: aflibercept
Drug: Brolucizumab-Dbll 120 MG/ML [Beovu] — Patients will be receiving intravitreal brolucizumab starting with 3 monthly doses followed by the treatment interval of 8 or 12 weeks based on the disease activity and BCVA.
  Other Names: Beovu
  Arms: brolucizumab
Drug: Ranibizumab 6 MG/ML [Lucentis] — Rescue therapy for patients with study drug related adverse events or with worsening of BCVA and OCT finding even on the shortest treatment interval when resistance to study drug is suspected.
  Other Names: Lucentis

SUMMARY:
This is a prospective randomised study comparing two intravitreal antiVEGF drugs - brolucizumab and aflibercept - in the treatment of retinal angiomatous proliferation (RAP). Patients with RAP confirmed on optical coherence tomography (OCT) and on OCT angiography (OCTA) will be randomised in two groups and followed for 52 weeks.

Patients in the first group will receive aflibercept - 3 injections monthly for the first 3 months and then in treat-and-extend regimen with minimal interval of 8 weeks and maximal interval of 16 weeks. Extension or shortening of the therapeutic interval will be possible in 2 or 4 week increments based on the visual acuity and disease activity assessed on OCT.

Patients in the second group will receive brolucizumab - 3 injections monthly in the first 3 months and then every 2 or 3 months based on the visual acuity and disease activity assessed on OCT.

Best corrected visual acuity (BCVA), central retinal thickness (CRT) on OCT and number of injections will be compared between both groups.

DETAILED DESCRIPTION:
Retinal angiomatous proliferation (RAP) is one of the variants of wet form of age-related macular degeneration (wAMD). Neovascularization in RAP grows from the retinal deep capillary plexus into the subretinal space where it forms subretinal and later choroidal neovascularization. It is often accompanied with high macular edema and pigment epithelium detachment (PED). As with other forms of wAMD, treatment with intravitreal antiVEGF drugs is highly effective. In our study, we would like to compare the efficacy of 2 antiVEGF drugs - aflibercept and brolucizumab - in the treatment of RAP.

This is a prospective, randomised, comparative study comparing the best corrected visual acuity (BCVA) and central retinal thickness (CRT) on optical coherence tomography (OCT) in the 16th, 26th and 52nd week of the study between patients with RAP treated with aflibercept and brolucizumab. In the 52nd week, the total number of injections between both groups will be also compared.

Visit plan:

Screening visit - 14 to 1 day prior to baseline. Informed consent will be signed prior to any other study procedures. Ocular and medical history will be written down. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT and OCTA of both eyes will be performed. Colour fundus photograph (FP) and red-free (RF) FP of the macula of both eyes will be performed. Based on the examination results, patients eligibility for the study will be assessed.

Baseline - day 1 - VFQ-25 questionnaire will be done with the patient. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. Based on the examination results, patients eligibility for the study will be assessed. Eligible patients will be randomised and study medication will be given.

Week 4, Week 8 - adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. Study medication will be given.

Week 16 - adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. OCTA of the study eye (SE) will be performed. Study medication will be given. Next treatment visit will be scheduled based on the disease activity on the OCT, the ocular examination findings and the BCVA:

1. group - aflibercept - treatment interval can be left on 8 weeks or extended by 2 or 4 weeks based on the presence or absence of subretinal or intraretinal fluid or PED on the OCT, on the BCVA and on the presence of other signs of disease activity on the fundus examination (e.g. haemorrhage, hard exudates). Final decision is on the investigator.
2. group - brolucizumab - aflibercept - treatment interval can be left on 8 weeks or prolonged to 12 weeks based on the presence or absence of subretinal or intraretinal fluid or PED on the OCT, on the BCVA and on the presence of other signs of disease activity on the fundus examination (e.g. haemorrhage, hard exudates). Final decision is on the investigator.

Week 24 to week 48 - adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. Study medication will be given. Next treatment visit will be scheduled based on the disease activity on the OCT, the ocular examination findings and the BCVA:

1. group - aflibercept - treatment interval can be extended or shortened by 2 or 4 weeks based on the presence or absence of subretinal or intraretinal fluid or PED on the OCT, on the BCVA and on the presence of other signs of disease activity on the fundus examination (e.g. haemorrhage, hard exudates). Maximal treatment interval can be 16 weeks, minimal 8 weeks. Final decision is on the investigator.
2. group - brolucizumab - aflibercept - treatment interval can be set to 8 or 12 weeks based on the presence or absence of subretinal or intraretinal fluid or PED on the OCT, on the BCVA and on the presence of other signs of disease activity on the fundus examination (e.g. haemorrhage, hard exudates). Final decision is on the investigator.

W26 - adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. OCTA of the study eye (SE) will be performed. Study medication will be given and next treatment visit will be scheduled based on the disease activity on the OCT, the ocular examination findings and the BCVA if planned based on patients treatment schedule.

W52 - VFQ-25 questionnaire will be done with the patient. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. OCTA of the study eye (SE) will be performed. Colour fundus photograph (FP) and red-free (RF) FP of the macula of both eyes will be performed.

Study procedures:

OCT - performed on Spectralis OCT (Heidelberg Engineering GmbH, Heidelberg, Germany). CRT will be assessed from automatic retinal thickness analysis in 9 ETDRS subfields including the central subfield. 49 horizontal scans in the angle of 20x20° 123 um apart in High resolution mode with noise reduction set to ART=4 will be performed.

OCTA - performed on Spectralis OCT (Heidelberg Engineering GmbH, Heidelberg, Germany). 512 horizontal scans in the angle of 20x20° 11 um apart in High speed mode with noise reduction set to ART=5 will be performed.

Disease activity assessment:

Based on the decision of the investigator. Shortening of the treatment interval is recommended when the BCVA decrease of more than 5 ETDRS letters is observed, in case of intra- or subretinal fluid or PED reappearance or increase on the OCT or when new haemorrhage or hard exudates are observed in the macula.

Extension of the treatment interval is recommended in the absence of intra- and subretinal fluid and PED on the OCT with better or stable BCVA, or in case the BCVA and OCT findings are stable after 3 injections in the shortest possible interval.

Rescue therapy:

Ranibizumab may be given as a rescue therapy in case of patients with study drug related sight threatening adverse events or with worsening of BCVA and OCT findings even on the shortest treatment interval when resistance to study drug is suspected. Switch to rescue therapy must be consulted with and approved by principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* age of 50 years or more at the time the informed consent is signed
* active RAP in the macula including fovea diagnosed on OCT and OCTA
* BCVA between 70 to 35 ETDRS letters (approx. 20/40 to 20/200 Snellen equivalent)
* decrease in BCVA caused primarily by the RAP in the study eye
* presence of intra- or subretinal fluid or PED in the central 1 mm of the macula on the OCT
* patient capable of signing the informed consent

Exclusion Criteria:

* other causes of choroidal neovascular membrane (CNV) than wAMD
* previous or current conditions of the study eye:

  1. subretinal haemorrhage comprising more than 25% of the lesion in the study eye
  2. scar or fibrosis comprising more than 50% of the lesion in the study eye
  3. presence of retinal pigment epithelium (RPE) tears or ruptures in the central 1 mm of the macula in the study eye
  4. total lesion size more than 8 papillary diameters (PD) as per OCT and FP examination
  5. uncontrolled glaucoma in the study eye defined as IOP of more than 25 mmHg despite the antiglaucoma treatment
  6. idiopathic or autoimmune uveitis in the study eye
  7. other pathologies in the macula of the study eye which can be expected to influence the BCVA (e.g. macular hole, retinal atrophy, epiretinal membrane, etc.)
  8. history of glaucoma surgery in the study eye or probability that it will be necessary in the future
  9. aphakia or pseudophakia with absence of the posterior lens capsule (with the exception of missing posterior capsule due to Nd:YAG laser capsulotomy) in the study eye
  10. myopia in the study eye with spherical equivalent of more than 8 dioptries before any refractive or cataract surgery
  11. significant opacities of the ocular media in the study eye including cataract, which can interfere with BCVA assessment or FP or OCT examination
  12. corneal transplantation or corneal dystrophy in the study eye
  13. irregular astigmatism or BCVA-lowering amblyopia in the study eye
  14. diabetic retinopathy, diabetic macular edema or any other retinal vascular disease in the study eye
  15. extraocular or periocular infection or inflammation (e.g. blepharitis, keratitis, conjunctivitis, scleritis, etc.) in any eye at the time of screening or baseline visit
  16. any intraocular infection or inflammation in any eye during 12 weeks (84 days) before the screening visit
  17. allergy or hypersensitivity to any component contained in the study drug
  18. pregnant or breastfeeding women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-04 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | Baseline and week 52
  BCVA change from baseline to week 52.
Central retinal thickness | Baseline and week 52
  CRT change from baseline to week 52.
Number of injections | Week 52
  Average number of injections per patient in each group.

SECONDARY OUTCOMES:
Dry macula | Week 52
  Number of patients without any intra- or subretinal fluid and PED on the OCT examination at week 52.
Significant visual gain | Week 52
  Number of patients who gained more than 15 ETDRS letters in each group.
Significant visual loss | Week 52
  Number of patients who lost more than 15 ETDRS letters in each group.
Adverse events | Week 52
  Number of drug or procedure related adverse events, such as uveitis, retinal breaks, intraocular haemorrhage etc.
Rescue | Week 52
  Number of patients who received rescue therapy in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pencak, M.D., Principal Investigator — Faculty Hospital Kralovske Vinohrady
Locations (1):
- Department of Ophthalmology, Faculty hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No